CLINICAL TRIAL: NCT05917912
Title: A Randomized, Double-blind, Placebo-controlled, 2-period, Crossover Study to Evaluate the Efficacy and Safety of ATX01 (Topical Amitriptyline Hydrochloride 15% w/w) in Adult Patients With Pain Due to Erythromelalgia (EM)
Brief Title: EASE (Efficacy of ATX01 Study in Erythromelalgia)
Acronym: EASE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AlgoTherapeutix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATX01-23-01-EM; 2022-003804-34 (EudraCT Number); 161942 (Other: IND)
Record Dates: First submitted 2023-06-05; First posted 2023-06-26 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2023-05

CONDITIONS: Erythromelalgia
MeSH Terms: conditions — Erythromelalgia | interventions — Amitriptyline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence A (Active Comparator): i)screening and randomization; ii) baseline period (3 weeks); iii) treatment period 1 with placebo(3 weeks); iv) wash-out period (3 weeks); v), treatment period 2 with ATX-01(3 weeks); vi) follow-up visit
  Interventions: Drug: Amitriptyline Hydrochloride; Drug: Placebo
- Sequence B (Active Comparator): i)screening and randomization; ii) baseline period (3 weeks); iii) treatment period 1 with ATX-01(3 weeks); iv) wash-out period (3 weeks); v), treatment period 2 with placebo (3 weeks); vi) follow-up visit
  Interventions: Drug: Amitriptyline Hydrochloride; Drug: Placebo

INTERVENTIONS:
Drug: Amitriptyline Hydrochloride — hydrogel bottle of ATX01 15% , 0,5ml (1pump) per hand, 1ml (2 pumps) per feet during 3 weeks
Drug: Placebo — hydrogel bottle of placebo , 0,5ml (1pump) per hand, 1ml (2 pumps) per feet during 3 weeks

SUMMARY:
The goal of this two-center, randomized, double-blinded, parallel-group, placebo-controlled clinical study is designed to compare the efficacy of twice daily applications of ATX01 versus placebo during two consecutive 3-week treatment periods. The primary objective is the comparison between Treatments (ATX01 15% vs. Placebo) of mean pain attack intensity score assessed for the final week of each treatment period using an 11-point Numerical Pain Rating Scale (NPRS). Mean pain attack intensity is defined as the sum of the pain intensity score of each pain attack during the last 7 full days (Day 14 to Day 20) of each Treatment Period divided by the total number of erythromelalgia pain attacks during that 7-day period.

Participants will apply on feet and/or hands twice a day in the morning and in the evening, approximately 12 hours apart from the morning administration for 3 consecutive weeks each and record the pain intensity of each attack that occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 years of age and older.
2. Documented diagnosis of erythromelalgia, as characterized by redness, warmth, and burning pain of the extremities (most commonly feet), typically precipitated by heat or exercise and relieved by cooling.
3. Mean pain attack intensity, measured on the 11-point NPRS, of ≥4 and ≤9 at baseline and ≥4 pain attacks per week as documented through eDiary use during the 3 weeks prior to randomization (Day -21 to Day -1).
4. Use of concomitant medications, with the exception of topical agents applied to the hands or feet, are permitted if the dose has been stable for at least 4 weeks preceding the screening visit and is planned to be maintained at the same regimen during the course of the study (prior treatment includes pharmacological and nonpharmacological treatments).
5. Patients having signed a written informed consent prior to any study related procedure.
6. Male patients should agree to use a condom along with another medically acceptable contraceptive method, where applicable according to local guidelines, if he is engaged in sexual activity with a woman of childbearing potential (WOCBP) from the day of the signature of the informed consent and up to 90 days after the end-of-study visit. Male patients should agree not to donate sperm until 90 calendar days after the last dose of study drug.
7. Females must comply with the following in order to be enrolled:

   1. WOCBP with negative pregnancy test results can be enrolled only if willing to use an acceptable contraceptive method, i.e. oral contraceptives, patch contraceptives, injection contraceptives, implantable hormonal contraceptives, male condom with intravaginal spermicide, diaphragm or cervical cap with spermicide, vaginal contraceptive ring, intrauterine device or system, surgical sterilization (hysterectomy, bilateral oophorectomy, and/or bilateral salpingectomy), tubal ligation/occlusion, vasectomized partner, or sexual abstinence, if this is the patient's current practice, from at least 14 days prior to the screening visit and throughout the study and for at least 30 days after the completion of the study.
   2. Or surgically sterilized for at least 6 months.
   3. Or menopausal, for at least 1 year.

Exclusion Criteria:

1. Clinical evidence of a pre-existing pain disorder in the extremities resulting from another cause than erythromelalgia, e.g. complex regional pain syndrome (CRPS), diabetic neuropathy, chemotherapy-induced peripheral neuropathy (CIPN).
2. Evidence of skin breakdown, ulcers, papules and > +2 pitting edema of the affected limbs.
3. Presence of glaucoma.
4. Presence of urinary retention (or significant prostatic hypertrophy at risk of urinary retention).
5. History of coronary artery disease.
6. History and /or presence of major depressive episode.
7. The patient has suicidal risk in the opinion of the investigator based upon clinical interview and the Columbia Suicide-Severity Rating Scale.
8. Pregnant or lactating women.
9. Abnormality in the 12-lead electrocardiogram (ECG) at screening that in the opinion of the investigator increases the risk of participating in the study, such as a corrected QT Fridericia (QTcF) interval >430 ms for males or >450 ms for females.
10. A history of additional risk factors for Torsade de Pointe (e.g. heart failure, hypokalemia, family history of Long QT Syndrome).
11. The use of concomitant medications within 24 weeks prior to Day 1 and/or during the study or the equivalent of 5 half-lives that prolong the QT/QTc interval, eg, Class 1 antiarrhythmics (e.g. quinidine, disopyramide, procainamide) and Class 3 antiarrhythmics (e.g. amiodarone, sotalol), antihistamines, antipsychotics known to prolong QT interval, and antimalarials (e.g. mefloquine, quinine), tricyclic antidepressants (e.g. AMT), tetracyclic antidepressants (e.g. maprotiline), cisapride.
12. The use of monoamine oxidase inhibitors within 24 weeks (or the equivalent of 5 half-lives) prior to Day 1 and/or during the study.
13. The use of opioids within 4 weeks (or the equivalent of 5 half-lives) prior to Day 1 and/or during the study.
14. History of illicit drug use or confirmed drugs of abuse at screening. Positive urine drug screen for prescribed medication is allowed at the discretion of the investigator.
15. Use of more than 2 analgesics (regardless of the route of administration) from different drug classes (including antidepressants and antiepileptics) on top of study drug.
16. Treatment with oral or topical amitriptyline or nortriptyline in the past 4 weeks or current treatment with any other tricyclic antidepressant.
17. Any known hypersensitivity to amitriptyline (regardless of the route of administration) in any salt form or to any constituent of the topical formulation.
18. Use of glutathione, vitamin E, minocycline, or calcium magnesium supplements within 12 weeks of screening.
19. Any topical treatment on treated extremities for any indication, other than cosmetic use of creams and lotions, within the 12 weeks prior to screening.
20. Any topical treatment for pain including use of:

    1. over-the-counter capsaicin on extremities within 12 weeks of screening,
    2. and/or Qutenza within 24 weeks of screening,
    3. and/or nonsteroidal anti-inflammatory drugs, menthol, methyl salicylate, local anesthetics within 1 week of screening.
21. Implanted active medical device (eg, spinal cord stimulator, intrathecal pump, or peripheral nerve stimulator) for the treatment of pain or any etiology.
22. Regional anesthetic block for pain of any etiology within 3 months prior to screening.
23. Intake in the 4 weeks preceding screening visit of any medication susceptible to inhibit or induce cytochrome P450 CYP2D6.
24. Poor metabolizers of CYP2D6 substrates.
25. Treatment with an investigational drug in the previous 4 weeks or greater, according to local requirements
26. Any condition that the investigator feels would place the patient at increased risk if the investigational therapy is initiated, such as, but not limited to, hyperthyroidism, convulsive disorder, advanced hepatic disease, pylorus, stenosis, or paralytic ileus.
27. The investigator considers the patient unfit for the study as a result of the medical interview, physical examination, or screening investigations, in particular any status or disease making the patient unable to follow instructions.
28. The patient is unable to apply the study drug on feet and/or hands.
29. The patient is an employee of the investigator, study site, sponsor, or contract research organization with direct involvement in the proposed study or other studies under the direction of the investigator, study site, or sponsor, or a family member of the site employee or the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Comparison between Treatments (ATX01 15% vs. Placebo) of mean pain attack intensity score | during the last 7 full days (Day 14 to Day 20) of each Treatment Period
  Comparison between Treatments (ATX01 15% vs. Placebo) of mean pain attack intensity score assessed for the final week of each treatment period using an 11-point Numerical Pain Rating Scale (NPRS). Mean pain attack intensity is defined as the sum of the pain intensity score of each pain attack during the last 7 full days (Day 14 to Day 20) of each Treatment Period divided by the total number of erythromelalgia pain attacks during that 7-day period

SECONDARY OUTCOMES:
Mean pain attack intensity score for complete treatment period | through study completion, an average of 15 weeks
  11 point Numeric Pain Rating Scale Scale: 0-10 10 means worst possible pain
Patient Global Impression of Change (PGI-C) score | through study completion, an average of 15 weeks
  Patient Global Impression: Global Change (PGI-C) Scale: 1-7 7 means very much worse
Change in pain interference with daily life using the Brief Pain Inventory - Short Form questionnaire (BPI-SF) | through study completion, an average of 15 weeks
  Brief Pain Inventory Pain Interference Questionnaire Scale: 0-10 10 means completely interferes
Change in quality of life, measured using the EuroQol-5-Dimension (EQ-5D) instrument | through study completion, an average of 15 weeks
  EuroQol-5-Dimension scale
Change in Beck Depression Inventory (BDI) score. | through study completion, an average of 15 weeks
  BDI Scale:0-3 3 means worse
Maximum pain intensity score, assessed by 11-point NPRS. | through study completion, an average of 15 weeks
  11 point Numeric Pain Rating Scale Scale: 0-10 10 means worst possible pain
Mean number of pain attacks per day | through study completion, an average of 15 weeks
Mean and maximum duration of pain attacks | through study completion, an average of 15 weeks
Mean frequency of use of rescue measures (e.g., cooling). | through study completion, an average of 15 weeks
Mean duration of use of rescue measures (e.g., cooling). | through study completion, an average of 15 weeks
Change in pain score before and after rescue measures (e.g., cooling). | through study completion, an average of 15 weeks
  11 point Numeric Pain Rating Scale Scale: 0-10 10 means worst possible pain

CONTACTS AND LOCATIONS:
Locations (2):
- Mayo Clinic, Rochester, Minnesota, United States
- Universitätsklinikum Erlangen Hautklinik, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No